CLINICAL TRIAL: NCT06924645
Title: Fecal Microbiota Transplantation for Preventing Gastrointestinal Symptoms in Extrapulmonary Neuroendocrine Neoplasms: A Real-World Study
Acronym: FMT-NENs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, caiwen, Chief Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0198
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-02

CONDITIONS: Treatment-related Gastrointestinal Toxicity (Including Diarrhea, Constipation, Nausea, and Vomiting); Extrapulmonary Neuroendocrine Neoplasms
MeSH Terms: conditions — Constipation; Nausea; Vomiting | interventions — Fecal Microbiota Transplantation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota transplantation (Experimental): Fecal Microbiota Transplantation (FMT) is delivered as a single dose of oral microbiota capsules within 72 hours before starting standard therapy.
  Interventions: Procedure: Fecal Microbiota Transplant (FMT)
- Control (Active Comparator): Standard Therapy Alone
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Procedure: Fecal Microbiota Transplant (FMT) — Fecal Microbiota Transplantation (FMT) is delivered as a single dose of oral microbiota capsules within 72 hours before starting standard therapy.
  Arms: Fecal microbiota transplantation
Other: Standard Therapy — Standard Therapy Alone
  Arms: Control

SUMMARY:
Existing studies have demonstrated that patients with different types of tumors exhibit significant increases in Enterobacter and Staphylococcus genera, along with marked decreases in Lactobacillus, Bacteroides, Bifidobacterium, and Enterococcus genera in their feces following chemotherapy. Research reports indicate a significant decline in bacterial diversity in rectal cancer patients post-chemotherapy, particularly showing reduced abundances of Porphyromonas, Peptostreptococcus, and Veillonella. Motoori et al. found that esophageal cancer patients undergoing combined chemotherapy with 5-FU, cisplatin, and docetaxel experienced significant reductions in intestinal Lactobacillus, alongside notable increases in Clostridium difficile and Enterococcus. Iida et al. confirmed that gut microbiota enhances the therapeutic efficacy of platinum-based agents and CpG oligonucleotides in cancer treatment. Concurrent studies suggest that probiotic supplementation during chemotherapy alleviates chemotherapy-related gastrointestinal reactions. Fecal microbiota transplantation (FMT), which involves transferring functional microbiota from healthy donors to patients' gastrointestinal tracts to reconstruct gut microbiota and improve microbial homeostasis, has emerged as a key clinical approach for regulating gut dysbiosis. It is currently recognized as the most effective established therapy for recurrent Clostridioides difficile infection (CDI). Previous studies have indicated FMT as a relatively safe, effective, and recommended treatment modality, while providing theoretical and experimental foundations for elucidating its efficacy and safety in preventing/reducing gastrointestinal symptoms associated with digestive tract cancer therapies.

This study aims to evaluate the improvement of treatment-related gastrointestinal symptoms and safety profile of FMT in extrapulmonary neuroendocrine tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender;
2. Anticipated survival period ≥3 months;
3. Pathologically confirmed diagnosis of extrapulmonary neuroendocrine neoplasms;
4. Development of gastrointestinal adverse reactions (including but not limited to diarrhea, constipation, vomiting, nausea, etc.) within three cycles of standard treatment;
5. Patients are capable and willing to sign an informed consent form and complete follow-up;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 1-3;
7. No use of oral/intravenous broad-spectrum antibiotics within 3 days prior to enrollment;
8. Ability to swallow capsules without chewing;
9. Adequate organ function confirmed by screening laboratory tests.

Exclusion Criteria:

1. Patients with major organ dysfunction or failure, including but not limited to cardiac insufficiency/heart failure, renal insufficiency/failure, or hepatic insufficiency/failure;
2. Uncontrolled or severe infection;
3. Known history of psychotropic drug abuse, alcoholism, or substance abuse;
4. Severe infection accompanied by sepsis or septicemia;
5. History of severe allergic reactions or known allergy to components of the liquid live bacterial enteric-coated capsules;
6. Female subjects with a positive pregnancy test, lactating women, or women of childbearing potential who refuse to use contraceptive measures during the observation period (15 weeks);
7. Patients with gastrointestinal perforation and/or fistula;
8. Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in treatment-related gastrointestinal symptoms | Assessed every two cycles (6 weeks)
  Hart Diarrhea Score

SECONDARY OUTCOMES:
Chemotherapy cycle delay rate | Assessed every two cycles (6 weeks)
Quality of Life (QoL) assessment | Assessed every two cycles (6 weeks)
  QOL assessment
Gut microbiota colonization | Assessed every two cycles (6 weeks)
  Performing 16S rRNA sequencing, metagenomic sequencing on the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China